CLINICAL TRIAL: NCT02949427
Title: The Oronasal Microbiota in Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ORIOME
Record Dates: First submitted 2016-10-20; First posted 2016-10-31 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Hematologic Malignancy; Bone Marrow Transplantation
Keywords: Microbiome; Mycobiome; Virome; Pediatric leukemia; Pediatric bone marrow transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The human microbiome is composed of unique groups of microorganisms occupying distinct habitats distributed throughout the human body. The Human Microbiome Project recently evaluated the bacterial composition of the microbiome in 18 (for women) and 15 (for men) body sites. Much initial attention in the field of microbiome research has focused on the bacterial contribution to a "healthy" microbiome. However, it is clear that other microorganisms, including fungi and viruses, are also distributed throughout the human body and serve as functional components of the microbiome.

The populations of microorganisms residing within the oral and nasal cavities make important contributions to human health and disease. These contributions may be especially important in immunosuppressed patients, including those patients receiving myelosuppressive chemotherapy or undergoing hematopoietic stem cell transplantation. In these patients, organisms typically considered as commensals can become pathogenic, either locally or systemically.

This observational study is primarily undertaken to evaluate the oral and nasal microbiota and to define the population of fungal organisms residing within the oral and nasal cavities in pediatric oncology patients before and after receiving protocol-directed chemotherapy and associated supportive care.

DETAILED DESCRIPTION:
Participants will be recruited from the patient population at the St. Jude Children's Research Hospital (SJCRH). Participants will be enrolled in the study according to their underlying primary diagnosis: acute myeloid leukemia (AML) and in patients undergoing hematopoietic stem cell transplantation (HSCT).

Patients will be asked to provide an oral wash and nasal swab sample at three time points during the course of their treatment at SJCRH. These samples will be used to characterize comprehensively the oronasal microbiota.

* Group 1 will include 30 patients with newly diagnosed AML. Within 72 hours of the start of chemotherapy, patients will provide an oral rinse and nasal swab sample. Participants will provide two subsequent oral rinse and nasal swab samples. The first (second total oral rinse and nasal swab sample) will be provided within 7 days of completion of "induction II" of therapy. The second (third total oral rinse and nasal swab sample) will be collected within 7 days of completion of therapy.
* Group 2 will include 30 allogeneic HSCT recipients. Prior to beginning their conditioning regimen, patients will provide an oral rinse and nasal swab sample. Participants will provide two subsequent oral rinse and nasal swab samples. The first (second total oral rinse and nasal swab sample) will be collected after completing their conditioning regimen on day +10 (plus or minus 7 days). The second (third total oral rinse and nasal swab sample) will be collected on day +30 (plus or minus 7 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 4 to 21 years.
* Group 1: Patients with newly confirmed diagnosis of acute myeloid leukemia (AML).
* Group 2: Patients scheduled to receive conditioning for allogeneic HSCT within 7 days.

Exclusion Criteria:

* Patients in group 1 who have received chemotherapy for more than 72 hours prior to enrollment (group 1) or started preparative regimen for allogenic stem cell transplant (group 2).
* Patients who are unable to perform the oral rinse or nasal swab collection procedure.
* Patients who have any condition that would place them at unnecessary risk secondary to providing oral and nasal samples.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent for study participation.

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children receiving care at SJCRH with new hematologic malignancies, as well as patients scheduled for HSCT, will be approached to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Diversity index of oronasal fungal microbiome (mycobiome) | Start of therapy through completion of therapy (up to 2 years)
  Diversity index is a measure of the richness of microbial species present in the sample. It is a single summary continuous numerical quantity for each sample.
Relative abundance of the oronasal fungal microbiome | Start of therapy through completion of therapy (up to 2 years)
  Relative abundance is percentage of each taxa of fungal, describing which fungal species are detected in a sample.

SECONDARY OUTCOMES:
Diversity index of oronasal bacterial microbiome | Start of therapy through completion of therapy (up to 2 years)
  Diversity index is a measure of the richness of microbial species present in the sample. It is a single summary continuous numerical quantity for each sample.
Relative abundance of the oronasal bacterial microbiome | Start of therapy through completion of therapy (up to 2 years)
  Relative abundance is percentage of each taxa of bacteria, describing which bacterial species are detected in a sample.
Diversity index of the oronasal viral microbiome | Start of therapy through completion of therapy (up to 2 years)
  Diversity index is a measure of the richness of microbial species present in the sample. It is a single summary continuous numerical quantity for each sample.
Relative abundance of the oronasal viral microbiome | Start of therapy through completion of therapy (up to 2 years)
  Relative abundance is percentage of each taxa of viruses, describing which viral species are detected in a sample.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Maron Alfaro, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols